CLINICAL TRIAL: NCT07184164
Title: Effect of Educational Program by Using Behavior Change Wheel Model on Knowledge, Behavior and Involvement in Substance Abuse Among Adolescents: A Quasi-experimental Study
Brief Title: Effect of Educational Program on Knowledge, Behavior and Involvement in Substance Abuse Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, Assistant Professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2/2023 FOR 11
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Substance Abuse Problem
Keywords: Adolescent; Alcohol and Drug Involvement; Behavior Change Wheel; Substance abuse; knowledge
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Educational Program by Using Behavior Change Wheel Model
  Interventions: Behavioral: Educational Program by Using Behavior Change Wheel Model
- Control Group (Active Comparator): Routine health education
  Interventions: Behavioral: Routine Health Education

INTERVENTIONS:
Behavioral: Educational Program by Using Behavior Change Wheel Model — The BCW model includes three layers: the behavior system, intervention functions, and policy categories, with the last not being applied in this study. The research was structured into four phases: assessment, planning, implementation, and evaluation.
  Phases of the Study Assessment Phase: Researchers introduced themselves to parents and adolescents through personal interviews, explaining the study's significance. They collected demographic data in the forensic and toxicology department, using various tools to assess adolescents' behaviors before the educational program.
  Planning Phase: A tailored BCW model encompassed a wide range of educational interventions. The content
  Arms: Study Group
Behavioral: Routine Health Education — Participants in the control group received the routine health education and advice from nurses and healthcare providers working in the study settings
  Arms: Control Group

SUMMARY:
The aim of study was to effect of educational program by using behavior change wheel model on knowledge, behavior and involvement in substance abuse among adolescents. The design of this study was a quasi-experimental design and the target population for the study was adolescents. Research hypothesis

- The application of an educational program based on behavior change wheel model has a positive impact on knowledge, behavior and involvement in substance abuse among adolescents.

DETAILED DESCRIPTION:
Substance abuse is of great concern to health issues worldwide, that typically initiated during adolescence, and it usually increases the likelihood of future physical, behavioral, social, and health issues. The Behavior Change Wheel can used as a practical and effective way of delivering real behavior change among adolescent's substance abuser. The aim of study was to effect of educational program by using behavior change wheel model on knowledge, behavior and involvement in substance abuse among adolescents. The design of this study was a quasi-experimental design and the target population for the study was adolescents. Total 226 samples were selected using the convenient sampling technique. Tool of the study consists of four tools which includes Tool I: An interviewing structured questionnaire sheet, Tool (II): Adolescents' behavior changes related to COM-B part of Behavior Change Wheel assessment form: Tool (III): Reported assessment checklist of the second part of Behavior Change Wheel, and Tool IV: Adolescent Alcohol and Drug Involvement Scale (AADIS).

ELIGIBILITY:
Inclusion Criteria:

* Ages between 10 and 18 years
* had no history of receiving prior educational program

Exclusion Criteria:

* Cardiac disease
* Pulmonary disease
* Liver function disorders
* Renal impairment
* Psychological disease

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 226 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Adolescents' behavior changes related to COM-B part of Behavior Change Wheel assessment form | 3 months
  This tool assesses adolescents' behavior changes related to substance abuse using the COM-B model (Capability, Opportunity, Motivation). It consists of 15 items measuring adolescents' feelings and experiences related to substance use. Scoring ranges from 0 to 30, with a cutoff of 60% (18 points) indicating satisfactory behavior change. Validity and reliability were established through expert review and a Cronbach's alpha greater than 0.80.
Reported assessment checklist of the second layer of Behavior Change Wheel | 3 months
  This checklist evaluates adolescents' knowledge and practices regarding substance abuse through two parts: knowledge assessment with 10 items and reported practices across nine intervention functions. Each section uses varying scoring systems with cutoff points at 60% for satisfactory performance. The tool's validity and reliability were confirmed by experts and a Cronbach's alpha above 0.81.
Adolescent Alcohol and Drug Involvement Scale (AADIS) | 3 Months
  The AADIS is a standardized self-report tool measuring adolescents' frequency of alcohol and drug use over the past month. It includes 14 items, where higher scores indicate greater substance use involvement. A cutoff score of 37 is used to identify potential substance use disorders based on DSM-IV criteria. Interpretations range from no use (0) to possible substance use disorder (37 or higher).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Shehata, Professor, Study Chair — Menoufia University
Locations (1):
- Menoufia University, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilchrist E, Johnson A, McMurran M, Stephens-Lewis D, Kirkpatrick S, Gardner B, Easton C, Gilchrist G. Using the Behaviour Change Wheel to design an intervention for partner abusive men in drug and alcohol treatment. Pilot Feasibility Stud. 2021 Oct 28;7(1):191. doi: 10.1186/s40814-021-00911-2. PMID 34711276
- [Background] Alarco-Rosales R, Sanchez-SanSegundo M, Ferrer-Cascales R, Albaladejo-Blazquez N, Lordan O, Zaragoza-Marti A. Effects of a School-Based Intervention for Preventing Substance Use among Adolescents at Risk of Academic Failure: A Pilot Study of the Reasoning and Rehabilitation V2 Program. Healthcare (Basel). 2021 Nov 1;9(11):1488. doi: 10.3390/healthcare9111488. PMID 34828534